CLINICAL TRIAL: NCT05000658
Title: Efficacy of Soluble Dexamethasone by Echo-guided Infiltration Through the Sacrococcygeal Hiatus in Refractory Sciatica: a Prospective Randomised Double-blind Study Versus Placebo
Brief Title: Efficacy of Soluble Dexamethasone in Refractory Sciatica
Acronym: Dexhia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC21_0148
Record Dates: First submitted 2021-08-04; First posted 2021-08-11 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Sciatica
Keywords: Reluctant Sciatica, Infiltrations, Soluble Dexamethasone
MeSH Terms: conditions — Sciatica | interventions — dexamethasone 21-phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): HSC one injection of 4 mL soluble Dexamethasone phosphate (16 mg) (equivalent to 100 mg Prednisone), followed by up to 16 mL saline (depending on tolerance)
  Interventions: Drug: Dexamethasone phosphate
- group B (Placebo Comparator): HSC one injection of 4mL of saline and then up to 16 mL of saline (depending on tolerance)
  Interventions: Drug: Dexamethasone phosphate

INTERVENTIONS:
Drug: Dexamethasone phosphate — HSC injection of 4mL

SUMMARY:
This is a phase 3 prospective randomised double-blind study versus placebo, measuring the efficacy of soluble Dexamethasone by echo-guided infiltrations through the sacro-coccygeal hiatus in intractable sciatica

DETAILED DESCRIPTION:
Injection of 4ml of Dexamethasone Phosphate Soluble or 4ml of saline solution depending on the randomisation arm

ELIGIBILITY:
Inclusion Criteria:

* Patients with sciatica of disc origin (radio-clinical concordance on MRI or CT) postero-lateral
* Duration of evolution greater than 3 weeks despite analgesic / AINS treatment, and less than 3 months
* EVA sciatica pain > 4/10
* Oswestry 30 at inclusion
* Patient aged 18 years and older
* Patient affiliated to a social security scheme
* Patient able to understand the protocol and having signed an informed consent
* Patient with an indication for corticosteroid infiltration in the context of their pathology

Criteria for non-inclusion

* Signs or risks of infection, in particular signs of virosis
* Poor local skin condition
* Anticoagulation with VKA or anti-Xa, or haemorrhagic disease
* Neurological deficit < 3/5 or signs of cauda equina irritation
* Tarlov's cyst or low dural sac below week 4
* Hypersensitivity to Lidocaine, Dexamethasone, or any of its excipients
* Infiltration of the spine within the previous 3 months
* Patient with bilateral sciatica
* Patient with sciatica of osteoarthritic origin
* Patients with chronic respiratory insufficiency
* Pregnant or breastfeeding women or women refusing effective contraception until M3
* Patient deprived of liberty or under legal protection (guardianship or curatorship)
* Patient under court protection
* Patients participating in another clinical research protocol involving a drug or medical device
* Patients unable to follow the protocol, as judged by the investigator
* Patient refusing to participate in the study
* Patient with clinically narrowed lumbar canal
* Patient with polyneuropathy or myelopathy
* Patient with sequelae of neuropathic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Effectiveness assessed by classical global algo-functional index: OSWESTRY | Week 3

SECONDARY OUTCOMES:
Value of Eva scale for evaluated effectiveness on lower back pain | Month 6
Value of Eva scale for evaluated effectiveness on lower back pain | Week 1
Value of Eva scale for evaluated effectiveness on lower back pain | Week 3
Value of Eva scale for evaluated effectiveness on lower back pain | Week 6
Value of Eva scale for evaluated effectiveness on lower back pain | Month 3
Value of Eva scale for evaluated effectiveness on sciatic pain | Week 1
Value of Eva scale for evaluated effectiveness on sciatic pain | Week 3
Value of Eva scale for evaluated effectiveness on sciatic pain | Week 6
Value of Eva scale for evaluated effectiveness on sciatic pain | Month 6
Number of days off work | Month 6
Value of score to scale Oswestry | Month 6
Value of score to scale Oswestry | Week 1
Value of score to scale Oswestry | Week 6
Value of score to scale Oswestry | Month 3
Value of score to SF36 self questionnaires | Month 6
Value of score to SF36 self questionnaires | Week 1
Value of score to SF36 self questionnaires | Week 3
Value of score to SF36 self questionnaires | Week 6
Value of score to SF36 self questionnaires | Month 3
Percentage of second injections required | Month 6
Number of patients undergoing secondary surgery | Month 6
Result of Clinical parameters | week 3
Result of Imaging parameters | week 3
Number of secondary effects | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Maugars, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No